CLINICAL TRIAL: NCT00210015
Title: A Multi-Center, Randomized, Parallel-Group, Double-Blind, Efficacy and Safety Study of INS37217 Nasal Spray Versus Placebo in Subjects With Perennial Allergic Rhinitis
Brief Title: A Study in Subjects With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-105
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

INTERVENTIONS:
Drug: INS37217 Nasal Spray

SUMMARY:
The purpose of this study was to determine the efficacy and safety of the study drug compared to placebo for the treatment of subjects with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented history of allergy to perennial allergens and demonstrated sensitivity by the results of prick or intradermal skin testing.
* Have a self-reported history of at least mild, intermittent rhinorrhea and nasal blockage/stuffiness due to allergies.
* Have not started or had a change in immunotherapy regimen.

Exclusion Criteria:

* Have a physical obstruction in the nose.
* Will likely have an acute increase in severity of allergic rhinitis due to seasonal aeroallergens during the trial.
* Have acute or chronic sinusitis or had previous sinus surgery resulting in a significant change in the sinus or nasal anatomy.
* Have rhinitis medicamentosa or any other acute or chronic condition that could confound evaluations of nasal symptoms.
* Have asthma of sufficient severity to require use of excluded medications.
* Have taken any medications excluded as listed in the protocol.
* Have a clinically significant acute or chronic disease or clinically significant laboratory abnormality.
* Are a current smoker, recent smoker or past smoker as defined in the protocol.

Age Groups: Child, Adult, Older Adult
Enrollment: 630
Dates: Start 2002-12; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
total nasal symptom score

SECONDARY OUTCOMES:
average total nasal symptom scores over various timepoints average individual symptom scores
global assessment of perennial allergic rhinitis symptoms
instantaneous assessment of symptoms
change from baseline in quality of life assessments
physical and anterior nasal exams
laboratory tests
ECG
vital signs
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, B.S.N., Study Director